CLINICAL TRIAL: NCT06021223
Title: Trial of a Chicken Extract for Improving Mental Energy and Mechanisms of Action in Healthy Adults: A Randomized, Double-blind, Placebo-controlled Exploratory Study
Brief Title: The Effects of Chicken Extract on Mental Energy in Healthy Adults and the Underlying Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brand's Suntory Asia (Industry)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEC-002
Record Dates: First submitted 2023-08-22; First posted 2023-09-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adults
Keywords: Mental energy; Chicken extract; Mechanisms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chicken extract supplement (high-dose) (Experimental): 140ml of chicken extract supplement (high-dose) to be consumed daily for 2 weeks
  Interventions: Dietary Supplement: Chicken extract supplement (high-dose)
- Chicken extract supplement (low-dose) (Experimental): 140ml of chicken extract supplement (low-dose) to be consumed daily for 2 weeks
  Interventions: Dietary Supplement: Chicken extract supplement (low-dose)
- Placebo (Placebo Comparator): 140ml of placebo (caesinate) to be consumed daily for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chicken extract supplement (high-dose) — 140ml of chicken extract supplement (high-dose) to be consumed daily for 2 weeks
  Arms: Chicken extract supplement (high-dose)
Dietary Supplement: Chicken extract supplement (low-dose) — 140ml of chicken extract supplement (low-dose) to be consumed daily for 2 weeks
  Arms: Chicken extract supplement (low-dose)
Other: Placebo — 140ml of placebo to be consumed daily for 2 weeks
  Arms: Placebo

SUMMARY:
This exploratory trial investigates the effect of a chicken extract supplement on mental energy and its potential underlying mechanisms of action among healthy adults using a randomized, double-blind, placebo-controlled clinical trial design. Mental energy is a multi-dimensional construct comprising transient feelings about fatigue, vigor and motivation and cognitive performance in terms of sustained attention and reaction time.

A sub-study investigates the immediate biochemical changes after taking chicken extract.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at 35-64 years of age
* Assessed by investigator to be in good health
* Normal cognition based on investigator's clinical judgement per the routine practice
* Modified PSQI score > 5
* Agree to participate in the study and provide written informed consent
* Agree to abstain from herbal extracts or dietary supplements throughout the study period

Exclusion Criteria:

* BMI < 18.5 or ≥ 27 kg/m2
* Concurrent pharmacological treatments
* Current systemic diseases or current/history of neurological or cerebrovascular diseases
* Active peptic ulcer, or a history of peptic ulcer within the last 2 years
* Medications or interventions in the last 4 weeks, which in the investigators' judgement could potentially affect the outcome measures
* Regular significant quantities of dietary supplements or herbal extracts (> 2 times a week) in the last 4 weeks
* Regular excessive caffeine consumption, heavy alcohol consumption or heavy habitual smokers
* Any drastic changes in lifestyle (including diet, smoking, sleep, exercise, and mental and physical activities) in the last 4 weeks
* Not able to maintain the same lifestyle throughout the study period
* Inadequate visual and auditory acuity to allow neuropsychological testing per investigator's judgment
* Inability to undergo fMRI scan
* Any consumption of chicken extract supplement, or carnosine or anserine supplement, in the preceding 4 weeks
* History of allergy to caseinate, milk, or chicken meat
* Women who are pregnant or lactating or intending to do so
* Current enrolment in another interventional study
* Subjects who show unstable sleep habits during the previous month
* Excessive blood donation or blood drawn prior to baseline

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Reaction time and sustained attention (composite) assessed by Cogstate Brief Battery (CBB) | At baseline and on Day 14
Reaction time assessed by Deary-Liewald reaction time task | At baseline and on Day 14
Sustained attention assessed by psychomotor vigilance test | At baseline and on Day 14
Sustained attention assessed by trail making test | At baseline and on Day 14
Fatigue assessed by Profile of Mood States (POMS) | Daily from baseline to Day 14
  POMS-fatigue scores range from 0 to 24, with higher score indicating greater fatigue.
Fatigue assessed by visual analogue scale (VAS) | Daily from baseline to Day 14
  VAS scores range from 0 to 100, with higher score indicating greater fatigue.
Vigor assessed by Profile of Mood States (POMS) | Daily from baseline to Day 14
  POMS-vigor scores range from 0 to 28, with the higher score indicating greater vigor.
Vigor assessed by visual analogue scale (VAS) | Daily from baseline to Day 14
  VAS scores range from 0 to 100, with higher score indicating greater vigor.
Motivation assessed by visual analogue scale (VAS) | Daily from baseline to Day 14
  VAS scores range from 0 to 100, with higher score indicating greater motivation.
Cerebral blood flow using arterial spin labelling magnetic resonance imaging (MRI) | At baseline and on Day 14
Cerebral oxygenation using functional MRI blood oxygenation level dependent (BOLD) imaging | At baseline and on Day 14
Whole body metabolic rate using indirect calorimetry | At baseline and on Day 14
  Resting body metabolic rate will be measured
Plasma global metabolome (metabolic profile) using liquid chromatography mass spectrometry (LCMS) | At baseline and on Day 14
  Plasma samples will be analyzed to putatively identify biomarkers of product intake by comparison of test group with control group using high-performance liquid chromatography coupled to mass spectrometer (LCMS). LCMS analysis allows the simultaneous and non-targeted analysis of a wide array of endogenous and exogenous metabolites.
Salivary cortisol level | At baseline and on Day 14
Plasma carnosine | At baseline and on Day 14
Plasma anserine | At baseline and on Day 14
Plasma L-histidine | At baseline and on Day 14
Plasma methylhistidine | At baseline and on Day 14
Plasma beta-alanine | At baseline and on Day 14

SECONDARY OUTCOMES:
Sleep quality measured by modified Pittsburgh Sleep Quality Index (PSQI) | At baseline and on Day 14
  In the PSQI, scores from the individual items are used to generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score, with a range of 0-21 points, with higher scores indicating poorer sleep quality. The modified PSQI measures the sleep quality in the past two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No